CLINICAL TRIAL: NCT04865445
Title: A Phase 1 Open-Label Study to Evaluate the Interaction Potential Between AT 527 and Midazolam in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Midazolam and AT-527 (R07496998)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-009
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AT-527 550 mg + midazolam (simultaneous) (Experimental): n=12
  Interventions: Drug: AT-527 550 mg + midazolam
- AT-527 mg + midazolam (staggered) (Experimental): n=12
  Interventions: Drug: AT-527 550 mg + midazolam

INTERVENTIONS:
Drug: AT-527 550 mg + midazolam — Day 1: 2 mg midazolam Day 3: 550 mg AT-527 and 2 mg midazolam in the morning and a second 550 mg AT-527 dose in the evening.
  Days 4 to 6: 550 mg AT-527 administered twice daily (BID) Day 7: 550 mg AT-527 and 2 mg midazolam in the morning and a second 550 mg AT-527 dose in the evening.
  Other Names: AT-527 is also know as R07496998
  Arms: AT-527 550 mg + midazolam (simultaneous)
Drug: AT-527 550 mg + midazolam — Day 1: 2 mg midazolam Day 3: 550 mg AT-527 and 2 mg midazolam (with dosing offset by 2 hrs) in the morning and a second 550 mg AT-527 dose in the evening.
  Days 4 to 6: 550 mg AT-527 administered twice daily (BID) Day 7: 550 mg AT-527 and 2 mg midazolam (with dosing offset by 2 hrs) in the morning and a second 550 mg AT-527 dose in the evening.
  Other Names: AT-527 is also know as R07496998
  Arms: AT-527 mg + midazolam (staggered)

SUMMARY:
Drug-drug interaction study of midazolam and AT-527 (R07496998)

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-29 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Concomitant use of prescription medications, or systemic over-the-counter medications
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of midazolam | Day 1, Day 3, Day 7
  Maximum plasma concentration (Cmax) and Area under the concentration-time curve (AUC)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AT-527 | Day 3, Day 7
  Maximum plasma concentration (Cmax) and Area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Montreal, Montreal, Quebec, Canada